CLINICAL TRIAL: NCT03559816
Title: Selective Use of Episiotomy: the Impact on Perineal Trauma. A Prospective Observational Study Based on a New Classification of Perineal Trauma.
Brief Title: Selective Use of Episiotomy: the Impact on Perineal Trauma.
Acronym: SEPT-1
Status: Completed | Type: Observational
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Simone Garzon, Principal Investigator, Universita di Verona
Other Study IDs: SEPT-1
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Perineal Tear; Episiotomy Wound; Delivery; Injury, Maternal
Keywords: Episiotomy; Vaginal delivery; Perineal trauma; Laceration; Classification of second-degree laceration
MeSH Terms: conditions — Wounds and Injuries; Lacerations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Selective use of Episiotomy: Vaginal delivery assisted with selective use of episiotomy and prospective classification of perineal laceration with a sub-classification of second-degree tears. Data of subclassifications are registered with data usually recorded in delivery ward register.
  Interventions: Other: Classification of perineal tears based on new classification; Procedure: Selective use of Episiotomy
- Not selective use of Episiotomy: Vaginal delivery assisted without a selective use of episiotomy. Data retrospectively retrieved by delivery ward register that were usually recorded.

INTERVENTIONS:
Other: Classification of perineal tears based on new classification — Classifications according to the American College of Obstetricians and Gynaecologists (ACOG) and the Royal College of Obstetricians and Gynaecologists (RCOG) and sub classification of second-degree lacerations based on the assumption that episiotomy involves the same anatomic structures of a second-degree laceration (perineal muscle, mucosa and skin), and divides them in two sub-groups, named A (if spontaneous vaginal tear is smaller than episiotomy) and B (if spontaneous vaginal tear is bigger than episiotomy).
  Groups: Selective use of Episiotomy
Procedure: Selective use of Episiotomy — Standardized selective use of Episiotomy as recommended by guidelines.
  Groups: Selective use of Episiotomy

SUMMARY:
Vaginal delivery is commonly accompanied by trauma of the genital tract. Perineal trauma is classified into four degrees based on anatomic structures involved and severity of lacerations according to the American College of Obstetricians and Gynaecologists (ACOG) and the Royal College of Obstetricians and Gynaecologists (RCOG). Episiotomy is an intentional perineal incision performed by midwifes or obstetricians to enlarge vaginal opening during the second stage of childbirth and has become the most common surgical procedure worldwide. A routine use of episiotomy was proposed to prevent severe spontaneous lacerations, although it failed to to demonstrate a clear protective role with no benefits both for mother and baby. Therefore the guidelines changed in a selective use of episiotomy, and we have introduced it in our routine obstetrics care. Nevertheless, second-degree lacerations comprise a wide range of lesions, from a minimal involvement to a massive damage of the perineal muscles. Therefore, it was never confirmed that selective use of episiotomy reduce the perianal trauma in the range of second degree lesions.

We designed a prospective observational study with the introduction of a new classification of perineal trauma recorded with the usual data retrieved in delivery ward register. The aim is to definitively investigate if selective use of episiotomy reduce the overall perineal trauma.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery

Exclusion Criteria:

* All situations in which episiotomy was recommended according to our Labour Ward's procedures (such as shoulder dystocia, breech presentation and operative delivery with vacuum) have been excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Unassisted vaginal delivery of the study period.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Overall Incidence of perineal trauma | At delivery
  Overall Incidence of perineal trauma
Incidence of different degree of perineal trauma | At delivery
  Incidence of different degree of perineal trauma
Incidence of different subgroup of second-degree perineal trauma | At delivery
  Incidence of different subgroup of second-degree perineal trauma based on new classification

CONTACTS AND LOCATIONS:
Overall Officials: Simone Garzon, M.D., Principal Investigator — Univerisity of Verona; Massimo Franchi, M.D., Principal Investigator — Univerisity of Verona; Francesca Parissone, M.D., Principal Investigator — Univerisity of Verona; Cecilia Lazzari, M.D., Principal Investigator — Univerisity of Verona; Antonio Simone Laganà, M.D., Principal Investigator — Università degli Studi dell'Insubria; Giovanni Zanconato, M.D., Principal Investigator — Universita di Verona; Ricciarda Raffaelli, M.D., Principal Investigator — Universita di Verona
Locations (1):
- AOUI Verona - University of Verona - Department of Obstetrics and Gynecology, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided